CLINICAL TRIAL: NCT00906204
Title: Prospective, Randomized, Double-Blind, Double-Dummy, Multicenter Trial to Assess Safety of Single Dose vs. Traditional Administration of Thymoglobulin Induction for Renal Transplantation
Brief Title: Safety Trial of Single Versus Multiple Dose Thymoglobulin Induction in Kidney Transplantation
Acronym: STAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wright State University (Other)
Collaborators: Sanofi (Industry); University of Arizona (Other); Wake Forest University (Other); University of Nebraska (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, R. Brian Stevens, MD, PhD, FACS, FAST, Professor of Surgery and Graduate Studies and Director, Transplantation Division, Wright State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 183-09-FB
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: End-Stage Renal Disease; Kidney Failure
Keywords: Renal transplantation; Kidney transplantation
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — thymoglobulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-dose Thymoglobulin (Experimental): Biological/Vaccine Single-dose rabbit Anti-thymocyte Globulin induction, 6 mg/kg IV infusion
  Interventions: Biological: Single-dose rabbit Anti-thymocyte Globulin induction
- Divided-dose Thymoglobulin (Active Comparator): Biological/Vaccine Divided-dose rabbit Anti-thymocyte Globulin induction, 1.5 mg/kg IV infusion QD x 4
  Interventions: Biological: Divided-dose rabbit Anti-thymocyte Globulin induction

INTERVENTIONS:
Biological: Single-dose rabbit Anti-thymocyte Globulin induction — 6 mg of rATG administered in a single dose on the day of kidney transplantation
  Other Names: Thymoglobulin; rATG
  Arms: Single-dose Thymoglobulin
Biological: Divided-dose rabbit Anti-thymocyte Globulin induction — 6 mg/kg total rabbit Anti-thymocyte Globulin dose administered as 1.5 mg/kg doses on 4 sequential days, beginning on the day of kidney transplantation.
  Other Names: Thymoglobulin; rATG
  Arms: Divided-dose Thymoglobulin

SUMMARY:
In a non-blinded pilot study conducted at the University of Nebraska Medical Center, evidence was found that a single large dose of Thymoglobulin on the day of kidney transplantation produced better kidney function than the standard dosing plan, when the same amount is divided into smaller doses on 4 days. This new study repeats that dose comparison, but with double-blinding and at multiple transplantation centers.

DETAILED DESCRIPTION:
This study is designed to confirm the one-year safety of single-dose rabbit anti-thymocyte globulin induction at kidney transplantation, compared to the conventional administration of the same overall dose divided into four smaller doses across four days. Two randomized groups of kidney transplant recipients will be each administered the drug Thymoglobulin according to a different dosing regimen. The control group will receive the usual and traditional regimen of a total of 6 mg/Kg divided into 4 doses, 1 on the day of transplantation and 1 each day on the next 3 days. The experimental group will receive the same total Thymoglobulin dose, 6 mg/Kg, but entirely on the day of transplantation.

The study will be double-blinded, with placebo doses of Thymoglobulin administered as needed to enrollees in the experimental group. Enrollment is targeted at 165, with 150 subjects needed to complete the study for adequate evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subject capable of giving written informed consent, with end-stage kidney disease, who is a suitable candidate for primary kidney transplantation
* Male or female subject who has reached legal age in the state where they reside and is at least 18 years of age
* Deceased or living donors
* Compatible ABO blood type
* Expanded-criteria donor (ECD) kidneys with a donor grade score of ≤ 25 (as developed by Nyberg, et al.)
* If Kidneys are pumped, they must meet the following pumping parameters: resistance <0.35 with a flow rate of >60 ml/min.

Exclusion Criteria:

* Recipient age >65 years
* PRA >50%, or donor-specific antibody
* CIT >30 hours
* Re-transplant patients
* Multi-organ transplant recipients (example: kidney/pancreas or kidney/liver)
* Renal transplant recipients planned for future pancreas transplantation
* Current unstable cardiovascular disease or history of myocardial infarction within the previous 6 months
* Current malignancy or history or malignancy (within the previous 5 years) with the exception of non-metastatic basal or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix that has been treated successfully.
* Hepatitis B and C recipients or active liver disease
* HIV positive recipients
* Primary disease requiring treatment with steroids after transplantation
* Expanded-criteria donor kidneys (current UNOS criteria) with a donor grade score of > 25
* Donation after cardiac death (DCD) donors
* Dual adult kidneys
* Recipients of pediatric (age <12 years) unilateral or en-bloc kidneys
* Previous treatment with rATG
* Known hypersensitivity, extensive exposure, or allergy to rabbits
* Pregnant
* Any condition that in the investigator's opinion may compromise study participation (e.g., history or likelihood of non-compliance with immunosuppression regimen, protocol visits, tests, and studies)

Relative Exclusion Criteria:

* Patients with a BMI > 37 should be considered on an individual basis based on overall health and body habitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R.Brian Stevens, MD, PhD, Principal Investigator — Wright State University, Dayton, Ohio
Locations (4):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Wake Forest University, Winston-Salem, North Carolina
  - The Methodist Hospital Research Institute, Houston, Texas

REFERENCES:
- [Background] Stevens RB, Mercer DF, Grant WJ, Freifeld AG, Lane JT, Groggel GC, Rigley TH, Nielsen KJ, Henning ME, Skorupa JY, Skorupa AJ, Christensen KA, Sandoz JP, Kellogg AM, Langnas AN, Wrenshall LE. Randomized trial of single-dose versus divided-dose rabbit anti-thymocyte globulin induction in renal transplantation: an interim report. Transplantation. 2008 May 27;85(10):1391-9. doi: 10.1097/TP.0b013e3181722fad. PMID 18497677
- [Background] Stevens RB, Foster KW, Miles CD, Lane JT, Kalil AC, Florescu DF, Sandoz JP, Rigley TH, Nielsen KJ, Skorupa JY, Kellogg AM, Malik T, Wrenshall LE. A randomized 2x2 factorial trial, part 1: single-dose rabbit antithymocyte globulin induction may improve renal transplantation outcomes. Transplantation. 2015 Jan;99(1):197-209. doi: 10.1097/TP.0000000000000250. PMID 25083614
- [Derived] Stevens RB, Wrenshall LE, Miles CD, Farney AC, Jie T, Sandoz JP, Rigley TH, Osama Gaber A. A Double-Blind, Double-Dummy, Flexible-Design Randomized Multicenter Trial: Early Safety of Single- Versus Divided-Dose Rabbit Anti-Thymocyte Globulin Induction in Renal Transplantation. Am J Transplant. 2016 Jun;16(6):1858-67. doi: 10.1111/ajt.13659. Epub 2016 Mar 7. PMID 26696251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial enrollment occurred between 3/30/2010 and 3/25/2014. Patients scheduled to undergo kidney transplantation were evaluated for trial suitability/enrollment in the transplant hospital or clinic just before transplantation, typically from a few hours to ~24 hours before transplantation.
Pre-assignment Details: Occasionally patients were evaluated and thought to be suitable trial candidates until transplantation was imminent, when they were ruled out by last-minute observation of medical problems or donor shortcomings.
Period: Primary Endpoint (Early Safety)
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin
Started | 45 | 52
Completed | 43 | 51
Not Completed | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Untransplantable donor kidney | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Secondary Endpoints (Long-term Safety)
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin
Started | 43 | 51
Completed | 41 | 48
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients who received a kidney transplant along with the study intervention, either single-dose or divided-dose rabbit anti-thymocyte globulin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin | Total
Number analyzed (Participants) | 44 | 51 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 48 | 90
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (11.8) | 49.0 (12.4) | 48.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 29 | 38 | 67
Region of Enrollment [Number; unit: participants]
  United States | 44 | 51 | 95
Type of kidney donor [Number; unit: participants]
  Living donor | 26 | 29 | 55
  Deceased donor | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint of 5 Components: Fever, Hypoxia, Hypotension, Cardiac Events, and Delayed Graft Function
Description: The composite endpoint components and definitions are:
  * Fever: Body temperature ≥ 38.5˚C.
  * Hypotension: After rATG initiation, systolic blood pressure ≤ 90 mmHg requiring de novo treatment with vasopressors.
  * Hypoxia: During transplantation surgery, increase in FiO2 to ≥ 60% following rATG initiation. Following transplantation, starting in recovery room, FiO2 ≥ 50% or nasal cannula delivering ≥ 3 liters, either singly or combined, for > 12 hours out of a 24 hour period.
  * Cardiac events: Myocardial Infarction, clinically significant dysrhythmia (atrial fibrillation, atrial flutter, ventricular fibrillation and ventricular tachycardia)
  * Delayed graft function (DGF): Requirement for dialysis within 7 days of transplantation
Time Frame: During first 7 days after kidney transplantation
Measure: Number; unit: participants
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin
Number analyzed (Participants) | 44 | 51
participants | 13 | 12
Statistical Analysis 1: Comparison: Single-dose Thymoglobulin vs Divided-dose Thymoglobulin; The analysis compares the rates at which patients in each of the two groups cumulatively exceed the five composite endpoint thresholds. There are five safety outcomes monitored during the first seven post-transplantation days. The rates of observed vs. possible safety outcomes are compared; Test type: Non-Inferiority or Equivalence — A one-sided alpha = 0.05, 85% power, an event rate of 0.70, equivalence margin of 0.20. Sample size = 75 patients per dose group, a total of 150 patients. Data analyzed will be counts of patients in each group who experience one or more component events of the primary endpoint during postoperative days one through seven. The DSMB requested an interim analysis after 80 patients and recommended ending the trial because the primary endpoint had been robustly reached; p = 0.64, Fisher Exact

2. Secondary Outcome: Patient Survival
Description: Kaplan-Meier estimate of the number of patients who survived for the 12 months after kidney transplantation.
Time Frame: 12 months post-transplantation
Measure: Number; unit: participants
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin
Number analyzed (Participants) | 44 | 51
participants | 44 | 50
Statistical Analysis 1: Comparison: Single-dose Thymoglobulin vs Divided-dose Thymoglobulin; Test type: Superiority or Other; p = 0.35, Log Rank

3. Secondary Outcome: Graft Survival
Description: Kaplan-Meier estimates of graft survival probability for 12 months after transplantation
Time Frame: 12 months post-transplantation
Measure: Number; unit: participants
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin
Number analyzed (Participants) | 44 | 51
participants | 42 | 50
Statistical Analysis 1: Comparison: Single-dose Thymoglobulin vs Divided-dose Thymoglobulin; Test type: Superiority or Other; p = 0.47, Log Rank

4. Secondary Outcome: Acute Kidney Rejection
Description: Kaplan-Meier probability estimates of rejection rates
Time Frame: 12 months post-transplantation
Measure: Number; unit: participants
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin
Number analyzed (Participants) | 44 | 51
participants | 5 | 5
Statistical Analysis 1: Comparison: Single-dose Thymoglobulin vs Divided-dose Thymoglobulin; Test type: Superiority or Other; p = 0.78, Log Rank

5. Secondary Outcome: Incomplete Thymoglobulin Infusion
Time Frame: First 7 days post-transplantation
Measure: Number; unit: participants
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin
Number analyzed (Participants) | 44 | 51
participants | 3 | 5
Statistical Analysis 1: Comparison: Single-dose Thymoglobulin vs Divided-dose Thymoglobulin; Test type: Superiority or Other; p = 0.72, Fisher Exact

6. Secondary Outcome: Kidney Function
Description: Estimated Glomerular Filtration Rate using the abbreviated MDRD formula (Modification of Diet in Renal Disease study)
Time Frame: 12 months post-transplantation
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin
Number analyzed (Participants) | 41 | 50
mL/min/1.73m^2 | 59.3 (15.6) | 61.3 (23.3)
Statistical Analysis 1: Comparison: Single-dose Thymoglobulin vs Divided-dose Thymoglobulin; Test type: Superiority or Other; p = 0.85, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: One year.
Description: Patient laboratory values and events were systematically collected on post-transplantation days 0 through 7, then on days 21, 42, 90, 180, 270, and 365. Review and collection of enrolled patient data was by specific clinical research nurse specialists at each study site withoverall review by a clinical trial Contract Research Organization.
Arm/Group | Single-dose Thymoglobulin | Divided-dose Thymoglobulin
Serious Adverse Events (participants affected / at risk) | 23/44 | 21/51
Other Adverse Events (participants affected / at risk) | 44/44 | 49/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-dose Thymoglobulin (N=44) | Divided-dose Thymoglobulin (N=51)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
serum sickness (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Atypical chest pain (Cardiac disorders) | 0 (0) | 1 (1)
hyperkalemia (Endocrine disorders) | 1 (1) | 2 (2)
abdominal fullness (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
death (General disorders) | 0 (0) | 1 (1)
orthostatic hypotension (General disorders) | 1 (1) | 0 (0)
cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
hepatitis C exposure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Leukopenia (Immune system disorders) | 0 (0) | 1 (1)
BK virus (Infections and infestations) | 1 (1) | 0 (0)
C. difficile (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Histoplasmosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Viral Gasteroenteritis (Infections and infestations) | 0 (0) | 2 (2)
rATG reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chronic lymphoid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Acute tubular necrosis (Renal and urinary disorders) | 2 (2) | 1 (1) — After post-transplantation day 7
Delayed graft function (Renal and urinary disorders) | 1 (1) | 1 (1)
Interstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Native nephrectomy (Renal and urinary disorders) | 1 (2) | 0 (0)
Nephrostomy tube placement (Renal and urinary disorders) | 0 (0) | 1 (1)
Perinephric hematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Rejection (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal vein thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wound hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-dose Thymoglobulin (N=44) | Divided-dose Thymoglobulin (N=51)
Anemia (Blood and lymphatic system disorders) | 14 | 14
Hemorrhage (Blood and lymphatic system disorders) | 3 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 14
Hypertension (Cardiac disorders) | 11 | 15
Hypotension (Cardiac disorders) | 4 | 5
Tachycardia (Cardiac disorders) | 5 | 2
Hyperglycemia (Endocrine disorders) | 18 | 21
Hyperkalemia (Endocrine disorders) | 8 | 12
Hyperparathyroidism (Endocrine disorders) | 0 | 3
Hyperphosphatemia (Endocrine disorders) | 5 | 7
Hypokalemia (Endocrine disorders) | 5 | 7
Hypomagnesemia (Endocrine disorders) | 15 | 12
Hypophosphatemia (Endocrine disorders) | 6 | 6
Osteopenia (Endocrine disorders) | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 4 | 7
Diarrhea (Gastrointestinal disorders) | 11 | 10
Gastric reflux (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 4 | 7
Edema (General disorders) | 4 | 9
Orthostatic hypotension (General disorders) | 2 | 4
Tacrolimus elevation/toxicity (General disorders) | 5 | 2
Elevated liver enzymes (Hepatobiliary disorders) | 2 | 4
Leukocytosis (Immune system disorders) | 3 | 10
Leukopenia (Immune system disorders) | 12 | 18
Neutropenia (Immune system disorders) | 1 | 3
BK virus (Infections and infestations) | 5 | 6
Pancytopenia (Immune system disorders) | 2 | 3
C. difficile (Infections and infestations) | 3 | 0
Respiratory infection (Infections and infestations) | 5 | 6 — Includes colds, sinusitis, bronchitis
Urinary tract infection (Infections and infestations) | 10 | 11
Possible rATG reaction (Injury, poisoning and procedural complications) | 2 | 6
Metabolic acidosis (Metabolism and nutrition disorders) | 7 | 7
Hyperlipidemia (Metabolism and nutrition disorders) | 7 | 2
Tremor (Nervous system disorders) | 0 | 5
Dysuria (Renal and urinary disorders) | 3 | 2
Elevated serum creatinine (Renal and urinary disorders) | 8 | 10
Proteinuria (Renal and urinary disorders) | 5 | 4
Rejection (Renal and urinary disorders) | 2 | 4
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Hernia (Surgical and medical procedures) | 3 | 1
Wound complication (Surgical and medical procedures) | 4 | 3 — Includes wound hematoma, seroma, drainage, slow healing

LIMITATIONS AND CAVEATS:
After an interim analysis at the trial mid-point, the trial was terminated because a futility trend analysis showed a >1.72% chance of the primary endpoint rates between the two groups achieving a significant difference with further enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No